CLINICAL TRIAL: NCT03375606
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous CSL730 in Healthy Caucasian and Japanese Subjects
Brief Title: Assessing the Safety and Tolerability of CSL730 in Healthy Caucasian and Japanese Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor decided to terminate this study in favor of development of subcutaneous administration.
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: CSL730_1001; 2017-003478-15 (EudraCT Number)
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSL730 (Experimental)
  Interventions: Biological: CSL730
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CSL730 — Solution for IV infusion
  Other Names: Recombinant trivalent human IgG1 Fc multimer
  Arms: CSL730
Other: Placebo — Saline solution for IV infusion
  Arms: Placebo

SUMMARY:
To assess the safety and tolerability of ascending doses of CSL730 after a single intravenous (IV) infusion in healthy Caucasian and Japanese subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females (postmenopausal or surgically sterile only) aged ≥ 20 to ≤ 55 years and of Caucasian or Japanese descent

Exclusion Criteria:

* Evidence of a clinically significant medical condition, disorder, or disease as judged by Investigator and / or study Medical Monitor.
* History of asthma (with the exception of childhood asthma that has resolved), chronic obstructive pulmonary disease, or recurrent or current respiratory infections; splenectomy; or recurrent or current gastrointestinal infections.
* Evidence of active or latent tuberculosis.
* Known or suspected hypersensitivity to the IP, to any excipients of the IP, humanized monoclonal antibodies, or Fc fusion protein therapeutics.
* History, or current diagnosis, of substance use disorder.
* Any abnormal clinical laboratory values deemed clinically significant by the Investigator and / or study Medical Monitor.
* Positive serology test result for human immunodeficiency virus antibody, hepatitis virus B surface antigen or hepatitis virus C antibody at Screening.
* Donation or loss of ≥ 480 mL of whole blood within 2 months or donation of plasma within 14 days before Day -1.
* Plans to participate in another investigational drug study while enrolled in this study, or has participated in any other investigational drug study in which they were known to have been administered a monoclonal antibody or biological IP within 4 months, any other investigational drug study within 60 days or > 3 investigational drug studies within 12 months before IP administration.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with adverse events overall, and by causality and severity | Up to 8 weeks after infusion

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of CSL730 in serum | Before study drug infusion and up to 56 days after the start of the infusion.
Area under the concentration-time curve from time 0 to the last collection time (AUC0-last) of CSL730 in serum | Before study drug infusion and up to 56 days after the start of the infusion.
Area under the concentration-time curve from time 0 extrapolated to time infinity (AUC0-inf) of CSL730 in serum | Before study drug infusion and up to 56 days after the start of the infusion.
Time of maximum observed concentration (Tmax) of CSL730 in serum | Before study drug infusion and up to 56 days after the start of the infusion.
Terminal elimination half-life (T1/2) of CSL730 in serum | Before study drug infusion and up to 56 days after the start of the infusion.
Total systemic clearance (CL) of CSL730 in serum | Before study drug infusion and up to 56 days after the start of the infusion.
Volume of distribution during the elimination phase (Vz) of CSL730 in serum | Before study drug infusion and up to 56 days after the start of the infusion.
Number of subjects with anti-CSL730 antibodies in serum | Before study drug infusion and up to 56 days after the start of the infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Study Director — CSL Behring
Locations (2):
- PRA Health Sciences, Groningen, Netherlands
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No